CLINICAL TRIAL: NCT05741346
Title: An Open-label Study to Evaluate the Long-term Safety of BCX9930 Monotherapy in Subjects With Paroxysmal Nocturnal Hemoglobinuria Who Previously Received BCX9930 in a BioCryst-sponsored Study
Brief Title: Long-term Safety of BCX9930 in Participants With Paroxysmal Nocturnal Hemoglobinuria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX9930-205; 2021-006776-17 (EudraCT Number)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: BCX9930; Factor D inhibitor; Proximal complement inhibitor; Oral therapy; Paroxysmal nocturnal hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BCX9930 (Experimental): Participants who had completed at least 12 weeks of treatment with BCX9930 in studies BCX9930-201, BCX9930-202, or BCX9930-203, and in the opinion of the investigator, had benefited from treatment with BCX9930 and were expected to continue benefiting from BCX9930, with no other effective treatment options, continued to receive BCX9930 tablets at a dose of 400 mg twice daily (BID) for up to 96 weeks. For participants who were permanently discontinuing BCX9930, in the absence of alternative complement inhibitor therapy, and if medically appropriate, the dose of BCX9930 was tapered based on investigator medical judgement.
  Interventions: Drug: BCX9930

INTERVENTIONS:
Drug: BCX9930 — Taken orally at 400 mg BID

SUMMARY:
This study was designed to provide continued access to BCX9930 for participants with Paroxysmal Nocturnal Hemoglobinuria (PNH) who had benefited from treatment with BCX9930 in another BioCryst-sponsored study for PNH who, in the opinion of the investigator, would benefit from continued treatment with BCX9930; who did not have access to other effective treatment options; and to monitor the safety of BCX9930 in participants continuing to receive BCX9930 for the treatment of PNH.

DETAILED DESCRIPTION:
This was an open-label, non-randomized study to evaluate the long-term safety of BCX9930 in participants with PNH. PNH is an acquired, rare, serious, and potentially life-threatening disorder characterized by destruction of red blood cells (RBCs) resulting from uncontrolled activity of complement.

The participants in this study had previously benefited from BCX9930 in BioCryst studies BCX9930-201, BCX9930-202, and BCX9930-203. As the development program was not being discontinued for safety reasons or due to a lack of efficacy, and the preliminary data available from the ongoing clinical studies in PNH did not change the current safety or efficacy profile for BCX9930, BioCryst remained committed to providing BCX9930 to those participants who had participated in the ongoing studies who were currently receiving benefit from BCX9930 and wished to continue treatment.

This study was used to meet that commitment by allowing for continued access to treatment with BCX9930 for any clinical study participant with PNH currently receiving treatment with BCX9930. As the development of BCX9930 was terminated, treatment was provided for a maximum of 96 weeks, as long as the investigator believed it was in the participant's best interest to continue treatment, or until the participant had access to alternative therapy for PNH, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female participants
* Were receiving treatment with BCX9930 in another clinical study of PNH and, in the opinion of the investigator, had benefited from treatment with BCX9930 and would have benefited from continued treatment with BCX9930, and who did not have access to other treatment options

Exclusion Criteria:

* Any clinically significant medical or psychiatric condition including alcohol or drug dependency that, in the opinion of the investigator or sponsor, would have interfered with the participant's ability to participate in the study or increased the risk of participation for that participant
* An ongoing adverse event, including a laboratory abnormality, or other unacceptable toxicity that, in the judgment of the investigator, compromised the ability of the participant to continue study-specific procedures or it was considered not to be in the participant's best interest to continue, or benefit-risk assessment was no longer in favor of the participant's continued treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Scheinberg, MD, PhD, Principal Investigator — Beneficência Portuguesa de São Paulo
Locations (11):
- Investigative Site, Paris, France
- Investigative Site, Budapest, Hungary
- Investigative Site, Ampang, Malaysia
- South Africa (3):
  - Investigative Site, Bloemfontein
  - Investigative Site, Cape Town
  - Investigative Site, Pretoria
- Investigative Site, Daejeon, South Korea
- Spain (2):
  - Investigative Site, Barcelona
  - Investigative Site, Valencia
- United Kingdom (2):
  - Investigative Site, Leeds
  - Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in France, Hungary, Malaysia, South Africa, South Korea, Spain, and the United Kingdom.
Pre-assignment Details: A total of 28 participants were enrolled. The participants were enrolled from previous studies BCX9930-201 (2020-000501-93), BCX9930-202 (2020-004438-39), or BCX9930-203 (2020-004403-14).
Groups:
- BCX9930: Participants who had completed at least 12 weeks of treatment with BCX9930 in studies BCX9930-201, BCX9930-202, or BCX9930-203, and in the opinion of the investigator, had benefited from treatment with BCX9930 and were expected to continue benefiting from BCX9930, with no other effective treatment options, continued to receive BCX9930 tablets at a dose of 400 milligram (mg) twice daily (BID) for up to 96 weeks. For participants who were permanently discontinuing BCX9930, in the absence of alternative complement inhibitor therapy, and if medically appropriate, the dose of BCX9930 was tapered based on investigator medical judgement.
Period: Overall Study
Arm/Group | BCX9930
Started | 28
Completed | 0
Not Completed | 28
Not completed — Withdrawn due to termination of study | 28

BASELINE CHARACTERISTICS:
Groups:
- BCX9930: Participants who had completed at least 12 weeks of treatment with BCX9930 in studies BCX9930-201, BCX9930-202, or BCX9930-203, and in the opinion of the investigator, had benefited from treatment with BCX9930 and were expected to continue benefiting from BCX9930, with no other effective treatment options, continued to receive BCX9930 tablets at a dose of 400 mg BID for up to 96 weeks. For participants who were permanently discontinuing BCX9930, in the absence of alternative complement inhibitor therapy, and if medically appropriate, the dose of BCX9930 was tapered based on investigator medical judgement.
Arm/Group | BCX9930
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0
  Ethnicity: Not Hispanic or Latino | 25
  Ethnicity: Not Reported | 1
  Ethnicity: Unknown | 2
  Race: American Indian or Alaska Native | 0
  Race: Asian | 5
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 13
  Race: White | 9
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant. No causal relationship with study intervention or with the clinical study itself is implied. An AE could be an unfavorable and unintended sign, symptom (including an abnormal laboratory finding), syndrome, or illness that developed or worsened during the clinical study. A serious adverse event (SAE) is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important event. An AE is considered treatment emergent if its start date was on or after the date of first dose of study treatment in Study 205 or if the AE was ongoing from the prior study. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: From Day 1 up to 30 days after last dose (up to approximately 100 weeks)
Population: Safety Population was defined as all participants who received at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930
Number analyzed (Participants) | 28
Participants | 27

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days after last dose (up to approximately 100 weeks)
Description: Safety Population was defined as all participants who received at least 1 dose of study intervention.
Arm/Group | BCX9930
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 16/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX9930 (N=28)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Intravascular haemolysis (Blood and lymphatic system disorders) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (6)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | BCX9930 (N=28)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1/13 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/13 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1/15 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Major depression (Psychiatric disorders) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Lung diffusion test decreased (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Dizziness (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 9 (15)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Splenomegaly (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Haemoglobinuria (Renal and urinary disorders) | 3 (5)
Haematuria (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Sterile pyuria (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (11)
Nasopharyngitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor decided to prematurely terminate the study due to business reasons. The decision to stop the development of BCX9930 was not due to safety reasons or due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT05741346/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05741346/SAP_001.pdf